CLINICAL TRIAL: NCT02696473
Title: Absorption of Naturally Present Compounds in Carrots and Their Appearance in Blood and Other Biofluids After Consumption (The Carrot Study)
Brief Title: The Bioavailability of Polyacetylenes From Carrots Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Carrot_01
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Bioavailability; Polyacetylenes; Falcarinol; Falcarindiol; Falcarindiol-3-acetate; Carrot; Biological Availability
MeSH Terms: interventions — Polyynes; falcarinol; falcarindiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Carrot Dose (Experimental): The volunteer will eat 250g carrot for breakfast with 2 slices of bread and 10g butter
  Interventions: Dietary Supplement: Carrot
- Low Carrot Dose (Experimental): The volunteer will eat 100g of carrot for breakfast with 2 slices of bread and 10g butter
  Interventions: Dietary Supplement: Carrot

INTERVENTIONS:
Dietary Supplement: Carrot
  Other Names: polyacetylene; falcarinol; falcarindiol; falcarindiol-3-acetate

SUMMARY:
Polyacetylenes, compounds found naturally in carrots, have shown promising anti-cancer and anti-inflammatory actions in vitro but have not been tested in vivo. To determine whether the polyacetylenes could have an effect in vivo, this study aims to determine whether they are detectible in human biofluids after the consumption of a portion of carrots and whether a difference is seen between a large and small portion.

DETAILED DESCRIPTION:
Volunteers will collect urine samples 24 hours prior to the 'test' day and a stool sample either the night before or the morning of the test session. They will have fasted blood taken before eating a portion of carrots with bread and butter. Further blood samples will be taken at 0.5, 1, 2, 3, 4, 6, 8 and 24 hours. All urine and all stool samples (after 4 hours) will be collected up to 48 hours after the carrot dose. They volunteers will attend two test sessions and will be randomised to receive high and low doses of carrot. At least a week will separate testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, BMI between 18.5 and 30

Exclusion Criteria:

* Metabolic or gastrointestinal conditions, allergies to carrot or bread, taking any medication that affects metabolism or digestion, smokers

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Detection of polyacetylene in biofluids | 72 hours
  The primary outcome will be whether a change in concentration of polyacetylene is seen between baseline and various time points in the biofluids after eating carrots.

SECONDARY OUTCOMES:
Detection of a difference between doses of polyacetylene in biofluids | 72 hours
  The secondary outcome will be whether there is a difference between the high and low dose concentrations of polyacetylenes at various time points after eating carrots.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Warner, Study Director — Newcastle University
Locations (1):
- Clinical Research Facility, Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No